CLINICAL TRIAL: NCT05317858
Title: A Randomized Pivotal Study Assessing the Safety and Efficacy of Targeted Blood-brain Barrier (BBB) Opening Using Exablate Focused Ultrasound During the Standard of Care Treatment of Brain Metastases of Non-small Cell Lung Cancer (NSCLC) Origin
Brief Title: Blood-brain Barrier (BBB) Opening Using Exablate Focused Ultrasound With Standard of Care Treatment of NSCLC Brain Mets
Acronym: LIMITLESS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BT012
Record Dates: First submitted 2022-03-01; First posted 2022-04-08 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Brain Tumor; Non Small Cell Lung Cancer
MeSH Terms: conditions — Brain Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; atezolizumab; cemiplimab; Nivolumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Imaging Core Lab is Blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- ICI Systemic Therapy with Exablate BBBO (Experimental): Using Exablate Model 4000 Type 2 for the treatment of NSCLC brain metastases in subjects who are undergoing planned ICI Systemic Therapy.
  Interventions: Device: Blood Brain Barrier Opening - Oncology; Drug: Pembrolizumab; Drug: Atezolizumab; Drug: Cemiplimab; Drug: Nivolumab; Drug: Iptilimumab
- Control Arm (ICI Systemic Therapy on-label use only) (Active Comparator): subjects will undergo planned on-label ICI Systemic Therapy.
  Interventions: Drug: Pembrolizumab; Drug: Atezolizumab; Drug: Cemiplimab; Drug: Nivolumab; Drug: Iptilimumab

INTERVENTIONS:
Device: Blood Brain Barrier Opening - Oncology — BBB opening via Exablate Type 2 system with microbubble resonators on the day of ICI infusion to treat brain metastases.
  Other Names: Exablate BBBO
  Arms: ICI Systemic Therapy with Exablate BBBO
Drug: Pembrolizumab — Pembrolizumab infusion
  Other Names: KEYTRUDA
Drug: Atezolizumab — Atezolizumab infusion
  Other Names: Tecentriq
Drug: Cemiplimab — Cemiplimab infusion
  Other Names: LIBTAYO
Drug: Nivolumab — Nivolumab infusion
Drug: Iptilimumab — Iptilimumab infusion

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of targeted blood brain barrier opening with Exablate Model 4000 Type 2.0/2.1 for the treatment of NSCLC brain metastases in patients who are undergoing planned FDA approved, on-label systemic therapy utilizing immune checkpoint inhibitors.

DETAILED DESCRIPTION:
This is a prospective, multi-center, randomized, two-arm, controlled, pivotal clinical trial to evaluate the safety and efficacy of targeted blood brain barrier opening using Exablate Model 4000 Type 2 for the treatment of NSCLC brain metastases in subjects who are undergoing planned FDA approved, on-label systemic therapy utilizing immune checkpoint inhibitors for their primary disease. The study will be conducted at up to 30 centers in the US. The immunotherapy regimen (every 3 weeks for 6 cycles) of prescribed ICI therapy is per the FDA approved labeling and the subjects prescribed standard of care therapy for their primary NSCLC. The study aims to demonstrate superiority of Exablate BBBO targeted to their brain metastases over the standard of care without Exablate BBBO with respect to the percentage of subjects achieving Objective Response Rate (ORR) by 6 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Participant is ≥ 18 years of age
* The participant provides written informed consent for the trial
* Participant is willing to comply with all study procedures for the duration of the study
* Participant has a Karnofsky Performance Status ≥ 70% and/or ECOG 0-2
* Participant is a NSCLC subject prescribed immune checkpoint inhibitor systemic therapy according to on-label use with the target brain lesion(s) measuring ≥ 0.5 cm in longest diameter. Target mets may include: De novo mets for which surgery and radiation can be deferred, Mets with or without history of prior radiation, Mets with history of radiation after at least 8 weeks since last radiation treatment, and In the event a previously treated met has progressed according to institutional practice within 4 weeks post radiation treatment, the met may be study eligible, and/or if in the opinion of the Investigator, the subject may benefit from the study procedure.
* Female subject is not planning pregnancy during the study duration and confirmed NOT PREGNANT each procedure day.
* Screening/Baseline laboratory values Screening/Baseline should adhere to local standard of care lab values for ICI therapy

Exclusion Criteria

* Participant has evidence of acute intracranial hemorrhage
* Participant at risk for spontaneous intracranial hemorrhage (e.g., history of metastatic melanoma or other tissue histology).
* Participant has signs and symptoms of increased intracranial pressure or symptomatic mass effect, midline shift or evidence of subfalcine, uncal or tonsillar herniation.
* Participant receiving Bevacizumab (Avastin) therapy, or other drugs with a proclivity for causing bleeding.
* History of bleeding disorders or tissue pathologies which increase the subject's risk of hemorrhage for anticoagulation medications, implement pre-surgical standard procedure to avoid increased risk of a bleeding event.
* Participant has an infectious viral infection such as active Hepatitis B, Hepatitis C or detectable HIV viral load or participants with active bacterial infection such as TB (Bacillus tuberculosis) that may, in the opinion of the investigator, interfere with the subject receiving the study therapy or procedures or otherwise impact their participation in the trial.
* Subjects with evidence of cranial or systemic infection.
* Participant has received a solid organ or hematopoietic stem cell transplant.
* Participant has received a live vaccine within 28 days prior to the first on-study ICI infusion with or without Exablate.
* Known sensitivity to DEFINITY® ultrasound contrast agent or hypersensitivity to perflutren microsphere or its components, e.g., polyethylene glycol, as found in MiraLAX and bowel prep products.
* Contraindications to MRI and gadolinium-DTPA including non-MRI-compatible implanted devices, severe claustrophobia, unable to lie supine in MRI.
* Subjects with significant liver dysfunction, (cirrhosis, hemochromatosis, severe alcohol abuse, or active hepatitis (autoimmune or infectious))
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first on-study ICI infusion with or without Exablate. Note: prophylactic steroid use for ICI and chemotherapy infusion per institutional practice is allowed per protocol.
* Has a known additional malignancy that requires active treatment that would interfere with study procedures.
* Known presence of leptomeningeal disease.
* Has a diagnosis of active autoimmune disease (e.g., autoimmune Hepatitis, Guillain-Barre Syndrome, etc.) requiring systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. History of (non-infectious) pneumonitis that requires steroids or has current pneumonitis
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Subject is currently enrolled in another intervention based clinical trial

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-08-12 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events | up to 6 months
  Adverse events [ Time Frame: Through study completion, up to 6 months]. All adverse events and/or Serious Adverse Events will be documented and reported according to CTCAE criteria.
tumor lesion(s) on the MRI images | up to 6 months
  Efficacy will be determined by the response of the tumor lesion(s) compared to baseline. Tumor lesions on the MRI images (units: mm) will be measured every three weeks up to six months.

SECONDARY OUTCOMES:
evaluation of Neuro Oncology Brain Mets (RANO-BM) response | up to 6 months
  The evaluation of the percentages of subjects that achieved the stable disease (SD), partial response (PR) as the best objective response using the response assessment in Neuro Oncology Brain Mets (RANO-BM) response criteria measured at baseline and every 3 weeks during each treatment cycle to up to 6 months of therapy.
Time to response for brain metastases by treatment arm [applicable to the completed stage 1a only] | up to 6 months
  The time to achieve a confirmed complete response or partial response for brain metastases by treatment arm as assessed using the RANO-BM criteria evaluated every 3 weeks up to 6 months during treatment cycles.

OTHER OUTCOMES:
Patient reported quality of life measurement questionnaires | up to 6 months
  patient reported health and quality of life questionnaire completed every 3 weeks up to 6 months during treatment cycle.
Measurement of BBB Opening | up to 6 months
  Measurement of blood brain barrier opening (BBBO) assessment of post-sonication contrast-enhanced MR imaging evaluated every 3 weeks up to 6 months in comparison with pre-sonication imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Manmeet Ahluwalia, MD, MBA, Principal Investigator — Miami Cancer Institute, Baptist Health South Florida
Locations (8):
- United States (6):
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Miami Cancer Institute at Baptist Health, Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - University of Maryland, Baltimore, Maryland
  - Rhode Island Hospital, Providence, Rhode Island
  - Johnston Willis Hospital, Richmond, Virginia
- Sunnybrook Research Institute, Toronto, Ontario, Canada
- Samsung Medical Center, Seoul, Seoul, South Korea